CLINICAL TRIAL: NCT04126824
Title: Prospective Randomized Controlled Clinical Trial: Superior Hypogastric Nerve Block for Pain Control After Uterine Artery Embolization: Effect of Addition of Steroids on Duration of Analgesia
Brief Title: Effect of Addition of Steroids on Duration of Analgesia
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jessica K. Stewart, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-001880
Record Dates: First submitted 2019-10-07; First posted 2019-10-15 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Uterine Fibroids; Adenomyosis
Keywords: Uterine Artery Embolization
MeSH Terms: conditions — Leiomyoma; Adenomyosis | interventions — Triamcinolone; Triamcinolone Acetonide; Bupivacaine; Iohexol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivacaine (Active Comparator): During the Uterine Artery Embolization (UAE) procedure, participants in this arm receive bupivacaine and contrast to enable visualization of the nerve block under fluoroscopy.
  Interventions: Drug: Bupivacaine; Other: Iohexol contrast
- Bupivacaine and Triamcinolone (Experimental): During the Uterine Artery Embolization (UAE) procedure, participants in this arm receive bupivacaine plus triamcinolone mixed with contrast to enable visualization of the nerve block under fluoroscopy.
  Interventions: Drug: Triamcinolone; Drug: Bupivacaine; Other: Iohexol contrast

INTERVENTIONS:
Drug: Triamcinolone — 40 mg triamcinolone administered as a Superior Hypogastric Nerve Block (SHNB)
  Other Names: Kenalog
  Arms: Bupivacaine and Triamcinolone
Drug: Bupivacaine — 0.5% bupivacaine (20 mL) administered as a Superior Hypogastric Nerve Block (SHNB).
  Other Names: Marcaine, Exparel
Other: Iohexol contrast — The appropriate amount of contrast to enable visualization of the nerve block under fluoroscopy given as a Superior Hypogastric Nerve Block (SHNB) will be administered.
  Other Names: Omnipaque

SUMMARY:
The purpose of the study is to investigate the differences in post-procedural pain scores and narcotic use among patients who receive a Superior Hypogastric Nerve Block (SHNB) with and without corticosteroid performed as part of the Uterine Artery Embolization (UAE) procedure.

DETAILED DESCRIPTION:
Investigators will enroll a total of 28 women undergoing the UAE procedure with 14 subjects in each study arm. This investigation is a single blind randomized control trial investigating the post-procedural analgesic effect of adding a corticosteroid (Triamcinolone) as an adjuvant to a SHNB that contains bupivacaine for patients undergoing UAE, compared to patients undergoing nerve block for pain control following UAE with local anesthetic only. Before and after the procedure, patients will be asked to complete online surveys in order to record their pain score (measured on the Visual Analog Pain Scale), opioid and other pain medication use, and other symptoms, such as nausea.

ELIGIBILITY:
Inclusion Criteria:

* females
* aged between 30 and 60 years
* diagnosed with symptomatic uterine fibroids and/or adenomyosis and scheduled to undergo UAE procedure

Exclusion Criteria:

* Contraindications to UAE
* SHNB is deemed unsafe for the patient
* Allergies to local anesthetic or steroid agent
* History of inflammatory bowel disease or ulcerative colitis
* Uncorrectable abnormal coagulation profile
* Diabetes mellitus

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2026-08-02 (Estimated); Study Completion 2027-08-02 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity Measure (mm) | Baseline, 240 hours
  The pain intensity is assessed using a visual analogue scale (VAS), which is a horizontal line 100 mm in length. Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain".

CONTACTS AND LOCATIONS:
Overall Officials: Jessica K Stewart, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California, Los Angeles, Westwood, Los Angeles, California
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No